CLINICAL TRIAL: NCT00960011
Title: Randomized Study of Self Gripping Semi-resorbable Mesh (PROGRIP) With Polypropylene Mesh in Open Inguinal Hernia Repair - the 6 Years Result
Brief Title: Comparative Study on Self-adhesive Mesh for Open Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Tung Wah Hospital (Other)
Responsible Party: Principal Investigator, Dr. Joe King-Man Fan, Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HERN-PROGRIP-01
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Hernia, Inguinal
Keywords: Inguinal hernia; mesh; progrip
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROGRIP (Experimental): Use of PROGRIP mesh for open inguinal hernia repair
  Interventions: Device: PROGRIP
- POLYPROPYLENE (Active Comparator): Use of Polypropylene mesh for open inguinal hernia repair
  Interventions: Device: POLYPROPYLENE

INTERVENTIONS:
Device: PROGRIP — Use of PROGRIP mesh for open inguinal hernia repair
  Other Names: PROGRIP MESH
  Arms: PROGRIP
Device: POLYPROPYLENE — Use of Polypropylene mesh in open inguinal hernia repair
  Other Names: Polypropylene mesh
  Arms: POLYPROPYLENE

SUMMARY:
Tension-less mesh repair is the most common procedure for inguinal hernia. Conventional heavy weight polypropylene meshes have been reported to stimulate inflammatory reaction and this is responsible for mesh shrinkage and postoperative chronic groin pain. Moreover, the fixation of the mesh with sutures is a tedious procedure and accounts for the majority of the operating time. A self gripping semi-absorbable mesh has been developed for anterior tension free inguinal hernia repair. It has the benefit of light weight property and does not require sutures for fixation. This study aims to compare the outcome of this self-gripping light weight mesh with the conventional heavy weight polypropylene mesh in inguinal hernia repair.

DETAILED DESCRIPTION:
Tension free mesh repair is the most common procedure for inguinal hernia repair. Conventional heavy weight polypropylene meshes have been reported to stimulate inflammatory reaction and this is responsible for mesh shrinkage when scar tissues are formed. In addition, the mesh requires fixation with sutures and there has been postulation that the fixation technique is related to postoperative chronic groin pain. Therefore, some authors have recommended the use of light-weight meshes and to limit the extent of fixation or to use non-compressive absorbable devices. In order to reduce the complications, a new self-gripping semi-resorbable mesh has been developed for anterior tension-free inguinal hernia repair.

The aim of this study is to compare the difference in operating time for open inguinal hernia repair with conventional prolene mesh and ProgripTM, which is a light-weight mesh with self-adhesive mechanism.

Methodology: Patients present with first episode of inguinal hernia are included into the study. Those with a sizable defect (>3cm defect), bilateral, inguino-scrotal hernia, irreducible, recurrence are excluded from study. Informed consents are signed before procedures and details of randomization are explained. Operations are performed by or under the supervision of specialist surgeons. Standardized inguinal dissection are performed. Randomization is carried out immediately before placement of mesh and after adequate inguinal dissection. PI / co-investigator phone to research assistant and ask for randomization result generated by computer. Total operative time, time from mesh placement to wound closure, blood loss, intra-operative complications, hospital stay, post-operative pain and analgesic used are documented.

Post-operative follow-up: Follow-up on day 14, 3 months, 6 months and 1 year post-op. Pain score, paraesthesia , chronic discomfort / pain, recurrence, seroma formation, testicular atrophy are documented. Thereafter, yearly follow-up is performed at clinic or by telephone to document the recurrence and chronic pain.

Parietene ProGrip™ (PP1208DR/ PP1208DL) Manufacturer: Sofradim Production Material: Monofilaments of polypropylene and polylactic acid (PLA) Color: Clear (undyed) Weight: 80g/m2 (before PLA resorbtion), 40g/m2 (after PLA resorbtion) Poresize: 1.7mm x 1mm

Material detailed description:

Parietene ProGrip™ is the first bio-component mesh comprised of monofilament polyester and a resorbable polylactic acid (PLA) gripping system which perfects true tension-free repair. The microhools cover the entire underside of the material allow complete anchoring of the mesh on the tissue. Self-gripping features also allows a strong and solid self-anchoring fixation and therefore making the hernia sac to fit perfectly to groin anatomy and move less underneath the prosthesis. Therefore, less suture is required and so operative time can be saved. Also less chance of nerve entrapment may cause low postoperative pain.

Surgipro Mesh (SPMM-35) Material: Monofilaments of polypropylene Color: Clear (undyed) Measurement: 15cmx15cm Thickness: 0.57mm

Description:

SURGIPRO Mesh is a non-absorbable, inert, sterile, porous surgical mesh knitted from mono-filament fibers of polypropylene polymer. The mesh exhibits high burst strength and tensile strength. The mesh is knitted in such fashion as to interconnect each mono-filament fiber and provide bi-dimensional elasticity while allowing the mesh to be cut to shape without unraveling.

Actions:

SURGIPRO Mesh is a porous, non-absorbable mesh used to repair or reinforce fascial defects following surgery or trauma and serves to provide additional support to such wounds during and following the wound healing period. Animal studies have shown that the polypropylene mono-filament fibers from which SURGIPRO Mesh is manufactured elicit a minimal acute inflammatory reaction in tissue, which is then followed by gradual encapsulation by fibrous tissue. In-growth of this fibrous tissue is permitted by the porosity of the knitted mesh structure. The mesh remains soft and pliable and the non-absorbable polypropylene fibers comprising the mesh resists loss of tensile strength in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and below 80
* Male or female patients
* Unilateral inguinal hernia
* First occurrence hernia

Exclusion Criteria:

* Inguino-scrotal hernia
* Recurrent inguinal hernia
* Incarcerated hernia
* Bilateral inguinal hernia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe KM Fan, MBBS MS FRCS, Principal Investigator — Department of Surgery, The University of Hong Kong
Locations (1):
- Department of Surgery, The University of Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Yes
upon email communication for identity verification
Supporting Information: Study Protocol
Time Frame: 5 years
Access Criteria: clinical researchers

REFERENCES:
- [Background] Chastan P. Tension-free open hernia repair using an innovative self-gripping semi-resorbable mesh. Hernia. 2009 Apr;13(2):137-42. doi: 10.1007/s10029-008-0451-4. Epub 2008 Nov 13. PMID 19005611
- [Background] Bringman S, Wollert S, Osterberg J, Smedberg S, Granlund H, Heikkinen TJ. Three-year results of a randomized clinical trial of lightweight or standard polypropylene mesh in Lichtenstein repair of primary inguinal hernia. Br J Surg. 2006 Sep;93(9):1056-9. doi: 10.1002/bjs.5403. PMID 16862613
- [Background] Helbling C, Schlumpf R. Sutureless Lichtenstein: first results of a prospective randomised clinical trial. Hernia. 2003 Jun;7(2):80-4. doi: 10.1007/s10029-002-0114-9. Epub 2003 Jan 30. PMID 12820029
- [Derived] Fan JKM, Yip J, Foo DCC, Lo OSH, Law WL. Randomized trial comparing self gripping semi re-absorbable mesh (PROGRIP) with polypropylene mesh in open inguinal hernioplasty: the 6 years result. Hernia. 2017 Feb;21(1):9-16. doi: 10.1007/s10029-016-1545-z. Epub 2016 Nov 26. PMID 27889845

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PROGRIP | POLYPROPYLENE
Started | 33 | 25
Completed | 22 | 23
Not Completed | 11 | 2
Not completed — Death | 5 | 0
Not completed — Lost to Follow-up | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROGRIP | POLYPROPYLENE | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (15.7) | 62.6 (16.0) | 62.3 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 18 | 22 | 40
Region of Enrollment [Number; unit: participants]
  Hong Kong | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Operating Time From Skin Incision to Wound Closure
Description: It measures the total operating time of 2 groups, measured from time started the skin incision to time finishing wound closure in terms of minutes.
Time Frame: Intra-operative record
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- PROGRIP(PG): It measures the total operating time of using PROGRIP mesh. it measured from time started the skin incision to time finishing wound closure in terms of minutes.
- POLYPROPYLENE(PL): It measures the total operating time of using POLYPROPYLENE mesh. it measured from time started the skin incision to time finishing wound closure in terms of minutes.
Arm/Group | PROGRIP(PG) | POLYPROPYLENE(PL)
Number analyzed (Participants) | 22 | 23
minutes | 39.2 (9.8) | 47.7 (7.6)

2. Secondary Outcome: Mesh Placement Time, Total Operative Time
Description: Time from mesh place to end of operation, and total time of operation
Time Frame: Intra-operative record
Measure: Mean (95% Confidence Interval); unit: Minutes
Groups:
- POLYPROPYLENE (PL): It measured from the time that the POLYPROPYLENE mesh is placed over inguinal canal for fixation to the time when operation finished in terms of minutes.
- PROGRIP (PG): It measured from the time that the PROGRIP mesh is placed over inguinal canal for fixation to the time when operation finished in terms of minutes.
Arm/Group | POLYPROPYLENE (PL) | PROGRIP (PG)
Number analyzed (Participants) | 23 | 22
Minutes
  Mesh placement time | 21 [14.8 to 27.2] | 11.8 [8.7 to 14.9]
  Total Operative time | 47.7 [39.7 to 55.7] | 39.2 [29.4 to 49]

3. Secondary Outcome: Seroma Formation at First Follow-up
Description: Seroma formation at first follow-up, go by clinical
Time Frame: 1 week after operation
Measure: Number; unit: number of patient with seroma at 1 week
Groups:
- PROGRIP; POLYPROPYLENE: Patient developed seroma clinically at 1 week after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
number of patient with seroma at 1 week | 5 | 8

4. Secondary Outcome: Overall Recurrence at 6 Years
Description: Overall recurrence at 6 years, including all recurrence
Time Frame: 6 years after operation
Measure: Number; unit: participants
Groups:
- PROGRIP; POLYPROPYLENE: Patient developed recurrence anytime from immediate post-op to 6 years after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
participants | 0 | 1

5. Secondary Outcome: Chronic Pain at 6 Years
Description: Patient with persistent chronic pain sensation at 6 years after operation. It described as painful sensation feeling around the operated site which is persistent and causing disturbance to daily normal life and attracted patients' attention.
Time Frame: 6 years after operation
Measure: Number; unit: participants
Groups:
- PROGRIP; POLYPROPYLENE: Patient with persistent chronic pain 6 years after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
participants | 3 | 3

6. Secondary Outcome: Patient With Testicular Atrophy From Post-op to 6 Years After Operation
Description: Patient with testicular atrophy from post-op to 6 years after operation, by clinical examination
Time Frame: 6 years after operations
Measure: Number; unit: participants
Groups:
- PROGRIP; POLYPROPYLENE: Patient with testicular atrophy from post-op to 6 years after operations
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
participants | 1 | 2

7. Secondary Outcome: Patient With Palpable Mesh at 6 Years After Operation
Description: Patient with clinical palpable mesh at 6 years after operation
Time Frame: 6 years after operation
Measure: Number; unit: participants
Groups:
- PROGRIP; POLYPROPYLENE: Patient with palpable mesh at 6 years after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
participants | 1 | 3

8. Secondary Outcome: Patient With Chronic Discomfort at 6 Years After Operation
Description: Patient with persistent chronic discomfort at 6 years after operation. It described as an unpleasant feeling around the operated site which is persistent and causing disturbance to daily normal life and attracted patients' attention. It is differentiate from pain sensation.
Time Frame: 6 years after operation
Measure: Number; unit: participants
Groups:
- PROGRIP; POLYPROPYLENE: Patient with chronic discomfort at 6 years after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
participants | 1 | 1

9. Secondary Outcome: Pain or Discomfort Affecting Daily Activities at 6 Years After Operation
Description: pain or discomfort which affecting daily activities at 6 years after operation
Time Frame: 6 years after operation
Measure: Number; unit: participants
Groups:
- PROGRIP; POLYPROPYLENE: pain or discomfort affecting daily activities at 6 years after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
participants | 1 | 0

10. Secondary Outcome: Total Number of Analgesic Used
Description: Total Number of Analgesic Used: Tablets
Time Frame: 1 week after operation
Measure: Mean (Standard Deviation); unit: Tablets
Groups:
- PROGRIP; POLYPROPYLENE: Total number of analgesic used at 1 week after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
Tablets | 10.4 (9.1) | 6.7 (8.2)

11. Secondary Outcome: Wound Pain at Rest at 1 Week After Operation
Description: Visual Analogue Score for measurement of wound pain at rest 1 week after operation
Time Frame: 1 week after operation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PROGRIP; POLYPROPYLENE: wound pain at rest at 1 week after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
score on a scale | 0.18 (0.39) | 0.13 (0.34)

12. Secondary Outcome: Wound Pain on Coughing at 1 Week After Operation
Description: wound pain on coughingt at 1 week after operation (Visual Analogue Score). It was in the form of 0-10 where 0 is no pain and 10 is maximal pain they experienced in their life. The higher the value, the more painful it is.
Time Frame: 1 week after operation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PROGRIP; POLYPROPYLENE: wound pain on coughing at 1 week after operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
score on a scale | 0.81 (0.5) | 0.83 (0.49)

13. Secondary Outcome: Post-operative Stay
Description: Post-operative stay (number of hours)
Time Frame: 1 week after operation
Measure: Mean (Standard Deviation); unit: hours
Groups:
- PROGRIP; POLYPROPYLENE: Post-operative stay (number of hours)
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
hours | 41.2 (40.5) | 28.6 (17.2)

14. Secondary Outcome: Days go Outdoor
Description: Post-op number of days that patient can go outdoor
Time Frame: 1 week after operation
Measure: Mean (Standard Deviation); unit: days
Groups:
- PROGRIP; POLYPROPYLENE: Days go outdoor
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
days | 2.5 (1.8) | 3.7 (2.7)

15. Secondary Outcome: Number of Participants Whose Response Was YES is Reported
Description: Patient will be asked by assessor in out-patient clinic about satisfaction about the whole arrangement of operation. We did not intend to grade the satisfaction but simply ask whether they are satisfied. Will be either YES or NO answer.
Time Frame: 1 week after operation
Measure: Number; unit: participants
Groups:
- PROGRIP; POLYPROPYLENE: satisfy with operation
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
participants | 20 | 23

16. Secondary Outcome: Size of Mesh (Longitudinal)
Description: Longitudinal size of mesh (in mm).
Time Frame: intra-operative record
Measure: Mean (Standard Deviation); unit: mm
Groups:
- PROGRIP; POLYPROPYLENE: size of mesh (longitudinal)
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
mm | 110.7 (7) | 106.7 (8.2)

17. Secondary Outcome: Size of Mesh (Vertical)
Description: Vertical size of mesh (in mm).
Time Frame: intra-operative record
Measure: Mean (Standard Deviation); unit: mm
Groups:
- PROGRIP; POLYPROPYLENE: size of mesh (vertical)
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
mm | 72 (6.7) | 66.7 (10)

18. Secondary Outcome: Wound Size
Description: Size of main wound
Time Frame: intra-operative record
Measure: Mean (Standard Deviation); unit: mm
Groups:
- PROGRIP: Size of skin wound using PROGRIP mesh for repair (in cm)
- POLYPROPYLENE: Size of skin wound using polypropylene mesh for repair (in cm)
Arm/Group | PROGRIP | POLYPROPYLENE
Number analyzed (Participants) | 22 | 23
mm | 50.7 (7.1) | 53.5 (5.7)

ADVERSE EVENTS:
Time Frame: from 2-6 years after operation
Description: unexpected operation unrelated mortality, Patients died of disease other than primary disease (hernia), nor due to treatment of such disease (hernia repair), nor due to material being used (mesh)
Arm/Group | PROGRIP | POLYPROPYLENE
Serious Adverse Events (participants affected / at risk) | 5/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROGRIP (N=22) | POLYPROPYLENE (N=23)
Non-surgery related mortality (Surgical and medical procedures) | 5 (5) | 0 (0) — Patients died of disease other than primary disease (hernia), nor due to treatment of such disease (hernia repair), nor due to material being used (mesh)

LIMITATIONS AND CAVEATS:
Small sample size. Up to 15% (5) patients died at 6 years after operation in progrip group. All deaths were not related to the primary disease (hernia), its treatment (hernia repair), nor material used (mesh).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes